CLINICAL TRIAL: NCT06570356
Title: Assessment of Depression Levels in Elderly Patients With an Orthopedic Fracture Compared to Patients After a Stroke.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shmuel Harofeh Hospital, Geriatric Medical Center (Other Government)
Responsible Party: Principal Investigator, Yochai Levy, Deputy Director, Shmuel Harofeh Hospital, Geriatric Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SH-101-22
Record Dates: First submitted 2024-08-20; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Depression; Old Age; Debility; Stroke; Fractures, Bone
MeSH Terms: conditions — Depression; Frailty; Stroke; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post stroke patients (Other)
  Interventions: Diagnostic Test: Geriatric Depression Scale - 15
- Post orthopedic fracture (Other)
  Interventions: Diagnostic Test: Geriatric Depression Scale - 15

INTERVENTIONS:
Diagnostic Test: Geriatric Depression Scale - 15 — a validated screening tool designed to identify depression in older adults. It consists of 15 simple yes/no questions that assess depressive symptoms.

SUMMARY:
Depression is common among elderly patients hospitalized due to acute conditions like strokes or osteoporotic fractures. It has significant impacts on quality of life, hospitalization rates, and mortality. Although studies have explored depression and its assessment, most focus on non-geriatric or ambulatory populations. This study examined depressive symptoms in elderly patients after a stroke or fracture. We assessed all patients for depression symptoms using the validated Geriatric Depression Scale - 15 item (GDS-15) and searched for contributing factors in each condition.

DETAILED DESCRIPTION:
Depression is a common condition among elderly patients hospitalized due to acute events and has both short-term and long-term prognostic impacts, including reduced quality of life, recurrent hospitalizations, and even mortality. Numerous studies have examined the effects of depression and the ability to assess it, but most have been conducted in non-geriatric populations and in ambulatory patients. It remains unclear whether different acute conditions are associated with distinct risk factors for depressive symptoms and whether depressive symptoms may have varying impacts across different acute conditions. In this study, we examined depressive symptoms in two groups of elderly patients-those with stroke and those with osteoporotic fractures. These are two common acute conditions in the geriatric population, both with significant implications for patient function and the incidence of depression.

Patients were recruited from a large geriatric hospital; all patients were capable of signing consent forms. At the beginning of their hospitalization, all patients will undergo a standardized depression screening test (GDS-15), and additional data will be collected from computerized medical records, including baseline data and the Functional Independence Measure (FIM) at the beginning and end of rehabilitation. Statistical analyses, including univariate analyses and multivariate regression, will be conducted to identify variables associated with depressive symptoms. Linear regression models will be constructed for each group based on the variables significantly associated with depression to assess the risk of depression according to the identified risk factors. To evaluate the risk of depression according to the models and assess the predicted GDS value's ability to classify participants with or without depression ROC curves will be used and AUC will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Age > 65 and hospitalization after stroke or fracture

Exclusion Criteria:

* Prior diagnosis of depression/current antidepressant treatment before hospitalization/ significant cognitive decline as indicated by a Mini-Mental State Examination (MMSE) score below 20/lacking the capacity to provide informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-02-02 (Actual); Primary Completion 2024-11-13 (Estimated); Study Completion 2024-11-13 (Estimated)

PRIMARY OUTCOMES:
Depression symptoms prevalence assessed by the Geriatric Depression Scale-15 | on recruitment and during hospitalization (avarege of about 14 days)
  Depression symptoms prevalence during hospitalization of patients after stroke or orthopedic fractures.

CONTACTS AND LOCATIONS:
Overall Officials: Yochai Levy, Principal Investigator — Tel Aviv University, Israel
Locations (1):
- Shmuel Harofe Geriatric Medical Center, Be’er Ya‘aqov, Israel

IPD SHARING:
Plan to Share IPD: No